CLINICAL TRIAL: NCT01280474
Title: Effects of Maternal Depressive Symptomatology on Pregnancy Outcomes and Newborn Development --- How is Paternal Psychopathology Involved?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Yi-Hua Chen, School of Public Health, Taipei Medical University
Other Study IDs: 99071
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Depression; Pregnancy
Keywords: depression during pregnancy; postpartum depression; pregnancy outcomes; newborn development; paternal psychopathology
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims at investigating the effects of maternal depressive symptomatology on pregnancy outcomes and newborn development. How paternal psychopathology is involved in the association will also be explored.

This is a three-year prospective cohort study. Three versions of questionnaires (the mother, the father, and the infant) will be developed first. For parents, data on self-reported symptomatology such as depression, anxiety, and stress will be collected, while for infants, maternal report on newborn development will be measured. Then, two medical centers and two regional hospitals will be selected. All pregnant women who undergo a first-trimester prenatal visit, who plan to carry the baby till term, and whose spouse is also willing to participate will be invited to join the study. The investigators expect to recruit a total of 194 pairs of depressive mothers and her spouses and 278 pairs of non-depressive mothers and her spouses in the study.

After the informed consent is obtained, one baseline assessment (i.e., the first trimester) and four follow-up assessments (i.e., the second trimester, the third trimester, one month postnatal and six months postnatal) will be implemented. Basically, prenatal investigation (for both mothers and fathers) will be carried out at the outpatient prenatal visit. Postnatal investigation (for the mothers, fathers and infants) will be processed at the pediatric outpatient visit when the infants are schedule for an immunization injection. After data are collected, descriptive, analytic and longitudinal data analyses will be performed to investigate the association between parental psychopathology and pregnancy outcomes and newborn development.

This study will explore the effects of the developmental trajectories of parental psychopathology on newborn growth during the critical stage of pregnancy. It is hoped that evidence based data could be obtained, examined, and applied in future prevention-intervention program to promote parental and newborn health, both physically and psychologically.

ELIGIBILITY:
Inclusion Criteria:

* Women who are pregnant within the gestational week of 14 (the first trimester) and have a prenatal visit at the selected hospitals.
* Women who expect to carry the baby to term.
* Women who are willing to provide information on their spouse or partner. And their spouse or partner also expresses the willingness to participate.

Exclusion Criteria:

* Pregnant women who are unable to provide information on their spouse or partner.
* Pregnant women's spouse or partner is unable to participate in this study.
* Pregnant women or their spouse or partner have difficulties in appropriately reading and completing a Chinese version questionnaire (e.g., illiteracy, not familiar with Chinese (e.g., foreign spouse), have major psychiatric illness, etc.)
* Women who are not appropriate to participate based upon doctoral or professional evaluation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and their spouses
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-08; Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hua Chen, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan